CLINICAL TRIAL: NCT02160600
Title: Role of Split Bolus Dual Energy Single Acquisition CT in Evaluation of Urological Diseases of the Upper Urinary Tract.
Brief Title: Dual Energy CT vs Standard Triple Phase CT-A Randomised Control Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, Dr.Dinesh Manoharan, Role of Split Bolus Dual Energy Single Acquisition CT in Evaluation of Urological Diseases of the Upper Urinary Tract., All India Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: IESC/T-457/29.11.2013
Record Dates: First submitted 2014-06-07; First posted 2014-06-10 (Estimated); Last update posted 2017-04-27 (Actual); Status verified 2017-04

CONDITIONS: Renal Cell Carcinoma; Renal Cysts; Transitional Cell Carcinoma; AML
MeSH Terms: conditions — Carcinoma, Renal Cell; Carcinoma, Transitional Cell

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- split bolus (Experimental): Patients will undergo diagnostic Split bolus DECT scan
  Interventions: Other: split bolus Dual energy CT
- Standard (Experimental): Patients will undergo routine multiphase diagnostic CT
  Interventions: Other: Standard multiphase CT

INTERVENTIONS:
Other: Standard multiphase CT
  Arms: Standard
Other: split bolus Dual energy CT
  Arms: split bolus

SUMMARY:
To compare SBDECT with standard Triple Phase Multi-Detector CT (TPMDCT) in renal mass evaluation in terms of appropriateness of treatment received after diagnosis. To determine SBDECT diagnostic accuracy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspected renal masses needing further evaluation with a contrast enhanced CT scan
* Patients who are referred for CT Urography

Exclusion Criteria:

* Patients not willing to participate in the study
* Age <18 yrs
* Pregnant females
* Patients with previous h/o serious allergic reactions or Contrast allergy
* Impaired renal function (estimated GFR<45mL/min/mm2)
* Sonographically proven benign renal mass needing no further evaluation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2014-04; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Appropriateness of the treatment recieved | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- All India Institute of Medical Sciences, New Delhi, National Capital Territory of Delhi, India